CLINICAL TRIAL: NCT02422017
Title: Topical Timolol Benefit in Venous Ulcers
Acronym: EETUV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2014_843_0022; 2014-005046-22 (EudraCT Number)
Record Dates: First submitted 2015-04-13; First posted 2015-04-21 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Venous Leg Ulcers
Keywords: Leg ulcer; wound; topical timolol
MeSH Terms: conditions — Leg Ulcer; Wounds and Injuries | interventions — Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Timolol (Experimental): Patients will receive one drop of timolol every 6cm ² every other day for twelve weeks in combination with dressings and compression.
  Interventions: Drug: Timolol; Other: Local care treatment
- Control (Other): Local care treatment only (dressing and compression applied every other day)
  Interventions: Other: Local care treatment

INTERVENTIONS:
Drug: Timolol — Patients will receive one drop of timolol every 6cm ² every other day for twelve weeks applied on the ulcer of interest
  Other Names: Timoptol
  Arms: Timolol
Other: Local care treatment — Local care treatment with dressing compression in accordance with standards applied every other day

SUMMARY:
Background: Venous Leg ulcers are a frequent pathology in dermatology and complex in their management. At the origin of high health costs and strong repercussions on quality of life for patients, they require long management and may be subject to possible complications.

In spite of appropriate treatment, 50-60% of these ulcers are not healed at 24 weeks.

Purpose: Topical beta adrenergic antagonists have shown efficacy in wound healing. The purpose of this study is to evaluate the efficacy and safety of treatment of chronic venous ulcers with topical timolol.

DETAILED DESCRIPTION:
Abstract: Complicating severe stages of chronic venous insufficiency, venous leg ulcers are common in dermatology and responsible for important health care costs. Healing remains long with many persistent cases after one year, despite compression and local dressings. Several pharmacological studies have demonstrated a benefit of beta-blockers on the wound healing process: present in the skin, the beta-adrenergic receptors play a role in wound healing. Their stimulation inhibits healing while blocking them promotes angiogenesis, fibroblast migration and keratinocyte migration. Using the topical timolol in several patients seems to confirm these effects: all ulcers treated with timolol healed in a few weeks whereas they did not evolve under local care and compression.

The purpose of this study is to demonstrate whether there is an interest in topical timolol for venous leg ulcers in combination with compression and wound dressings versus placebo. The primary endpoint is to evaluate the healing rate to W12. The effects will be evaluated with photography, evaluation of the surface of the ulcer at W12 compared to W0. The research of side effects will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to a social security scheme patients
* Informed consent
* Patients over 18 years
* Ulcer lasting for at least 24 weeks with no improvement observed after 4 weeks of well conducted treatment (compression and local care)
* Presence of one or more venous leg ulcers (objectified by a Doppler ultrasound dated within 6 months and ABPI ≥ 0.8)
* Ulcers with a surface of 5 to 50 cm ² and at granulation stage
* Study ulcer must be at least 2 cm from Any Other ulcer on same extremity.
* If several ulcers present, the greatest is selected
* Granulation tissue ≥ 50%

Exclusion Criteria:

* Minors under guardianship, deprived of liberty, not looking at treatment, lack of signed consent, pregnant women, demented patients
* Ulcer lasting for less than 24 weeks
* Granulation tissue <50%
* Obliterative arteritis (ABPI <0.8)
* Infection of the ulcer (need to treat the infection before any inclusion criteria be compatible)
* Non-cardioselective beta-blocker treatment
* Bradycardiac treatment
* Patients under diltiazem, verapamil (calcium antagonists)
* Reaching underlying noble structures, tumor acutisation wound
* Immunosuppression
* Diabetes unbalanced (HbA1c> 8%)
* Severe Malnutrition (albumin <25g / L)
* Anemia <10g/dl
* Contraindication to beta-blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Success rate | 12 weeks
  Assess the healing rate in patients treated with topical timolol associated with wound dressing and compression for 12 weeks, compared to patients treated with wound dressing and compression.
  Success is defined as an ulcer surface relative reduction >= 40%

SECONDARY OUTCOMES:
Complete healing | 12 weeks
  Complete healing of the ulcer i.e. 100% regression of the ulcer surface and replaced by an epidermised tissue.
Tolerance (cardiac-related serious adverse events) | 12 weeks
  To assess local and cardiac safety of timolol by cardiac-related serious adverse events evaluation
Quality of life evolution | Baseline and 12 weeks
  Evaluation of the quality of life of patients by the Dermatology Life Quality Index (DLQI) scale at baseline and after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

REFERENCES:
- [Result] Baltazard T, Senet P, Momar D, Picard C, Joachim C, Adas A, Lok C, Chaby G. Evaluation of timolol maleate gel for management of hard-to-heal chronic venous leg ulcers. Phase II randomised-controlled study. Ann Dermatol Venereol. 2021 Dec;148(4):228-232. doi: 10.1016/j.annder.2020.11.009. Epub 2021 Feb 4. PMID 33551214